CLINICAL TRIAL: NCT05792735
Title: A Prospective, Open-Label, Single-Arm and Multicentre Phase II Study to Explore the Efficacy and Safety of Neoadjuvant Cadonilimab Plus Chemotherapy Following Short-Course Radiotherapy in Middle and Lower Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Cadonilimab Plus Chemotherapy Following Short-Course Radiotherapy in Locally Advanced Rectal Cancer
Acronym: NeoCaCRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Wan He, Professor Wan He, Shenzhen People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shenzhen CRC-004
Record Dates: First submitted 2023-02-09; First posted 2023-03-31 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Rectal Carcinoma
Keywords: Anti-CTLA-4/PD-1 bispecific antibody; Neoadjuvant chemotherapy; Rectal cancer; Short-course radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Consolidation Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cadonilimab group (Experimental): Cadonilimab is administrated with 6mg/kg and repeated every 2 weeks.
  Interventions: Drug: Cadonilimab Injection; Radiation: Short-course radiotherapy; Drug: Consolidation chemotherapy

INTERVENTIONS:
Drug: Cadonilimab Injection — Cadonilimab, an anti-CTLA-4/PD-1 bispecific antibody, at a dose of 6mg/kg is given in combination with chemotherapy every 2 weeks preoperatively and postoperatively.
  Other Names: AK104
Radiation: Short-course radiotherapy — Preoperative short-course radiotherapy (5x5 Gy)
  Other Names: SCRT
Drug: Consolidation chemotherapy — Oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil bolus 400 mg/m2 on day 1, and 5-fluorouracil infusion 2400 mg/m2 for 48 h) every 2 weeks for total 6 cycles preoperatively and postoperatively.
  Other Names: mFOLFOX6

SUMMARY:
The goal of this clinical trial is to test the efficacy and safety in patients with locally advanced middle and lower rectal cancer. The main questions it aims to answer are:• Whether Cadonilimab combined with chemotherapy following short-course radiation can improve pathological complete response(pCR) rate? •Are the toxicities of the combination therapy manageable? Participants will be given radiation of 5 Gy for 5 days and then neoadjuvant Cadonilimab combined with modified fluorouracil, leucovorin, and oxaliplatin (mFOLFOX6) for 6 cycles. Without progressed disease, total mesorectal excision (TME) or transanal local excision will be performed. If clinical complete response was received, watch and wait strategy is one of choices. Adjuvant Cadonilimab plus mFOLFOX6 for another 6 cycles could be suggested for non-pCR participants,while surveillance is also suitable for pCR ones.

DETAILED DESCRIPTION:
Long-term synchronous chemoradiation (CRT) with sequential TME is the treatment recommended by current guidelines for locally advanced rectal cancer (LARC). The latest STELLAR study showed that preoperative short-course radiotherapy (SCRT) combined with preoperative chemotherapy is safe and effective and can be used as an alternative to conventional CRT in LARC [1]. In recent years, new therapies blocking immune checkpoints (cytotoxic T lymphocyte-associated molecular protein 4 (CTLA-4), programmed cell death 1 (PD1) and programmed cell death ligand 1 (PD-L1)) have achieved landmark achievements in the field of cancer therapy. Several clinical trials are evaluating the efficacy of a combination of RT and immune checkpoint inhibitors (ICIs) in rectal cancer (NCT02948348, NCT04124601, NCT04558684). The results of the study suggest that radioimmunotherapy is safe and effective in rectal cancer. A number of studies have shown that combined PD-1 and CTLA-4 blockade is associated with a higher response rate whereas more toxicities in multiple tumor types. Cadonilimab is a tetrameric PD-1/CTLA-4 bispecific antibody, based on the Akeso Tetrabody platform. It introduces novel T cell targeting mechanisms of action that may provide an improved therapeutic index and a favorable toxicity profile compared to PD-1 and CTLA-4 combination therapy. The study of SCRT combined with Cadonilimab and chemotherapy in middle and lower LARC has not been reported at home or abroad.

Therefore, this study plans to recruit 27 patients with middle and lower LARC to explore the efficacy and safety of radiation of 5 Gy for 5 days followed by Cadonilimab 6mg/kg plus mFOLFOX6 (oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil bolus 400 mg/m2 on day 1, and 5-fluorouracil infusion 2400 mg/m2 for 48 h) every 2 weeks for total 6 cycles preoperatively. The primary endpoint is the pathological complete response (pCR) after surgery. The secondary endpoints consist of a clinical complete response (cCR), major pathological response (MPR), objective response rate (ORR), recurrence-free survival (RFS), overall survival (OS) and safety. Clinical response was evaluated by endoscopy, digital rectal examination and pelvic MRI. Safety was analyzed in all patients who receive at least one dose of treatment. The exploratory endpoint covers the quality of life.

After surgery, non-pCR patients receive adjuvant Cadonilimab combined with mFOLFOX6 for 6 cycles while pCR ones have two options: adjuvant treatment which is the same as the neoadjuvant regimen or observation. As for cCR patients, TME or transanal local excision is one of options while the watch and wait (W&W) strategy can also be considered especially for ultra-low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 yeas and ≤79 years. The gender is not limited.
2. Histopathology confirmed the diagnosis of rectal adenocarcinoma.
3. Patients with rectal cancer based on endoscopic ultrasound and / or pelvic MRI contrast + contrast, chest CT, head MRI or CT + contrast, or positron emission tomography / computed tomography （PET / CT）, staging criteria per American Joint Committee on Cancer (AJCC) 8th edition cancer stage, cT 3-T4 / N + M0.
4. At least 20 unstained sections of formalin-fixed paraffin-embedded tumor tissue sections, or fresh tumor tissue, can be provided for genomic and proteomic testing.
5. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0- 1.
6. Adequate bone marrow and organ function meets the following criteria:

   1. Neutrophil count (ANC)≥1.5×l09/L
   2. Platelet (PLT) ≥80×109/L
   3. Hemoglobin (Hb) level ≥90 g/L
   4. Total bilirubin level≤1.5×ULN
   5. Alanine aminotransferase (ALT) level≤3×ULN
   6. Aspartate aminotransferase (AST) level ≤3×ULN
   7. International normalized value (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5×ULN
   8. Serum creatinine (Cr) level ≤1.5×ULN
   9. Creatinine clearance #50 ml/min (Calculated according to the Cockcroft-Gault formula)

Exclusion Criteria:

1. Previous history of severe hypersensitivity to other monoclonal antibodies or any component of Cadonilimab.
2. Preoperative pathology was diagnosed as squamous cell carcinoma or neuroendocrine tumor
3. Within 5 years before enrollment for malignancies other than colorectal cancer with negligible risk of metastasis or death (e. g., expected 5-year OS> 90%) and expected radical results after treatment (e. g., adequately treated cervical carcinoma in situ, basal or squamous cell skin carcinoma, localized prostate carcinoma for curative intent, ductal carcinoma in situ surgically treated with curative intent).
4. Previous treatment against the PD-1 receptor or its ligand PD-L1 or the cytotoxic T lymphocyte-associated protein-4 (CTLA-4) receptor.
5. History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, series, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis related to antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, vasculitis, or glomerulonephritis; patients with autoimmune-related hypothyroidism were eligible for stable-dose thyroid hormone replacement therapy; patients with type 1 diabetes under control after a stable insulin regimen were eligible to participate in this study;
6. Usage of systemic immune activation drugs (including but not limited to interferon or Interleukin-2) within 4 weeks prior to enrollment or within 5 half-lives of the drug (whichever is shorter);
7. Usage of systemic corticosteroids (> 10 mg/d of prednisone equivalent) or other systemic immunosuppressive agents (including but not limited to prednisone, prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents [anti-TNF]) within 2 weeks prior to enrollment. Local, ocular, intra-articular, nasal, and inhaled corticosteroids are permitted;
8. Patients requiring baseline and subsequent MRI tumor evaluation with previous allergic reactions to intravenous contrast agents may use preventive steroids;
9. Allowing the use of inhaled corticosteroids for chronic obstructive pulmonary disease, corticosteroid hydrochloride (e. g., fluorohydrocortisone) in patients with orthostatic hypotension, and low-dose corticosteroid maintenance for adrenal cortical insufficiency.
10. Patients with previous allogeneic bone marrow transplantation or previous solid organ transplantation.
11. Idiopathic pulmonary fibrosis, drug-induced pneumonia, mechanical pneumonia (i. e. bronchiolitis obliterans), history of idiopathic pneumonia or chest CT scan at screening showed evidence of active pneumonia.
12. Any live vaccine (e. g., vaccine against infectious diseases, such as influenza vaccine, varicella vaccine, etc.) within 4 weeks (28 days) before enrollment.13 Active infections, including tuberculosis (TB) (clinical diagnosis including clinical history, physical examination and imaging findings, and TB tests performed per local medical practice), hepatitis B {known HBV surface antigen (HBsAg) positive and HBVDNA 1000 cps / ml}, hepatitis C or human immunodeficiency virus (HIV antibody positive).
13. Patients with prior or cured HBV infection (defined as hepatitis B core antibody positive and HBsAg negative) were to be eligible to participate in the study only if HBVDNA was negative (HBVDNA˂ 1000 cps / ml);
14. Patients with positive hepatitis C (HCV) antibody are not eligible for the study only if polymerase chain reaction shows negative HCVRNA;
15. Clinically meaningful basic medicine, disease (e. g., dyspnea, pneumonia, pancreatitis, poorly controlled, poorly controlled diabetes, infection active or poorly controlled, or drug or alcohol abuse).
16. Presence of severe neurological or psychiatric disorders, including dementia and epileptic seizures.
17. The NCI-CTCAE grade 2 peripheral neuropathy.
18. Female patients during pregnancy or lactation.
19. Chronic bowel disease or short bowel syndrome.
20. Dihydropyrimidine dehydrogenase (DPD) enzyme deficiency.
21. Major cardiovascular diseases, such as New York Heart Association heart disease (grade II or higher), myocardial infarction within 3 months before randomization, unstable arrhythmia, or unstable angina pectoris.
22. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must have an optimized stable medical regimen as determined by the treating physician, consulting a cardiologist if required.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response Rate | Up to 6 months
  The proportion of patients with no tumor cells in the postoperative specimens

SECONDARY OUTCOMES:
Disease Free Survival Time from the date of treatment administration until the date of the first documented event of: disease recurrence Disease Free Survival | Up to 5 years
  Time from the date of treatment administration until the date of the first documented event of: disease recurrence following surgery (preferably biopsy proven), or death - whichever occurs first
Overall Survival | Up to 5 years
  Overall survival is defined as time from the date of treatment administration until the date of death from any cause.
Objective Response Rate | Up to 6 months
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
Clinical Complete Response | Up to 6 months
  Digital examination of rectum and multi-point puncture of colonoscopy indicate no tumor, and ultrasound colonoscopy and tumor markers
  and MRI are normal, which is considered as clinical complete response.
Major Pathological Response Rate (MPR) | Up to 6 months
  The proportion of cancer cells in the resected tumors and lymph nodes is less than 10%.
Number of participants with treatment-related adverse events (TRAE) as assessed by CTCAE v5.0 | Up to 6 months
  Number of patients with AE, TRAE, immune-related AE (irAE), serious adverse event (SAE) assessed by CTCAE v5.0, change from baseline in liver function, kidney function, peripheral blood counts, etc. at 3 months

OTHER OUTCOMES:
Quality of life (QoL) | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated using the European O-rganization for Reasearch and Treatment of Cancer Quality of Life Questionnaire-C30（EORTC QLQ-C30） (range 0-100). It evaluates the quality of life from 30 aspects, including appetite, mental status, sleep quality, fatigue, etc. The higher scores mean a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Jin J, Tang Y, Hu C, Jiang LM, Jiang J, Li N, Liu WY, Chen SL, Li S, Lu NN, Cai Y, Li YH, Zhu Y, Cheng GH, Zhang HY, Wang X, Zhu SY, Wang J, Li GF, Yang JL, Zhang K, Chi Y, Yang L, Zhou HT, Zhou AP, Zou SM, Fang H, Wang SL, Zhang HZ, Wang XS, Wei LC, Wang WL, Liu SX, Gao YH, Li YX. Multicenter, Randomized, Phase III Trial of Short-Term Radiotherapy Plus Chemotherapy Versus Long-Term Chemoradiotherapy in Locally Advanced Rectal Cancer (STELLAR). J Clin Oncol. 2022 May 20;40(15):1681-1692. doi: 10.1200/JCO.21.01667. Epub 2022 Mar 9. PMID 35263150
- [Background] Hodi FS, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Cowey CL, Lao CD, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hill A, Hogg D, Marquez-Rodas I, Jiang J, Rizzo J, Larkin J, Wolchok JD. Nivolumab plus ipilimumab or nivolumab alone versus ipilimumab alone in advanced melanoma (CheckMate 067): 4-year outcomes of a multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1480-1492. doi: 10.1016/S1470-2045(18)30700-9. Epub 2018 Oct 22. PMID 30361170
- [Background] Sharma P, Siefker-Radtke A, de Braud F, Basso U, Calvo E, Bono P, Morse MA, Ascierto PA, Lopez-Martin J, Brossart P, Rohrberg K, Mellado B, Fischer BS, Meadows-Shropshire S, Abdel Saci, Callahan MK, Rosenberg J. Nivolumab Alone and With Ipilimumab in Previously Treated Metastatic Urothelial Carcinoma: CheckMate 032 Nivolumab 1 mg/kg Plus Ipilimumab 3 mg/kg Expansion Cohort Results. J Clin Oncol. 2019 Jul 1;37(19):1608-1616. doi: 10.1200/JCO.19.00538. Epub 2019 May 17. PMID 31100038
- [Background] Shamseddine A, Zeidan YH, El Husseini Z, Kreidieh M, Al Darazi M, Turfa R, Kattan J, Khalifeh I, Mukherji D, Temraz S, Alqasem K, Amarin R, Al Awabdeh T, Deeba S, Jamali F, Mohamad I, Elkhaldi M, Daoud F, Al Masri M, Dabous A, Hushki A, Jaber O, Charafeddine M, Geara F. Efficacy and safety-in analysis of short-course radiation followed by mFOLFOX-6 plus avelumab for locally advanced rectal adenocarcinoma. Radiat Oncol. 2020 Oct 7;15(1):233. doi: 10.1186/s13014-020-01673-6. PMID 33028346